CLINICAL TRIAL: NCT02831803
Title: A Pilot Study to Evaluate the Feasibility of Walnut and Extra Virgin Olive Oil Supplementation in Older Adults Being Treated for Hypertension
Brief Title: Nuts and Extra Virgin Olive Oil Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: California Walnut Growers Association (Unknown); C.H.O. American, Natural and Organic Olive Oil Producer Association (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00028877
Record Dates: First submitted 2016-07-11; First posted 2016-07-13 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): All participants will receive an 8-week supply of walnuts and Extra Virgin Olive Oil (EVOO). Study supplements will consist of 28 gm of walnuts and 32 gm of EVOO per day. Participants will be instructed how to consume the proper amount of walnuts and EVOO and to report their consumption using a compliance diary. The walnuts are pre-packaged in daily servings (one 28 g packet per day) and measuring spoons will be provided with the olive oil to assist participants in consuming it appropriately. Participants will also receive recipes and other written information that will assist them in incorporating both the nuts and olive oil into their existing dietary patterns.
  Interventions: Dietary Supplement: Walnuts; Dietary Supplement: Extra Virgin Olive Oil

INTERVENTIONS:
Dietary Supplement: Walnuts — 28 gm/day in single-serve package
Dietary Supplement: Extra Virgin Olive Oil — 32 gm/day provided in 3, 34 ounce bottles

SUMMARY:
This study is designed to test the feasibility of asking older adults with high blood pressure to supplement their daily diets with walnuts and extra-virgin olive oil.

DETAILED DESCRIPTION:
Even though cardiovascular disease (CVD) continues to be the leading cause of death in the United States, Americans have yet to widely adopt evidence-based dietary modifications necessary to reduce CVD risk factors. Encouraging evidence from the Prevención con Dieta Mediterránea (PREDIMED) trial indicates that adding olive oil and nuts to the diets of older adults in Spain substantially impacted CVD risk factors and events.

A large trial testing EVOO and nuts in a U.S. population is needed to determine if supplementing with EVOO and nuts can reduce risk of cardiovascular events and mortality in adults living in the U.S. Prior to launching a large trial, it is important to assess whether adults 55 and older would be interested in participating in a supplementation trial such as PREDIMED. Additionally, it is important to assess if they are willing to consume the nuts and EVOO and attend study related-data collection visits.

ELIGIBILITY:
Inclusion Criteria:

* Being treated for hypertension-defined by being prescribed at least one hypertension medication; willing to comply with study visits, as outlined in the protocol; able to read and speak English; no allergies or hypersensitivities to olive oil or nuts; ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Plans to move from the study area in the next 8 weeks; dementia that is medically documented or suspected; homebound for medical reasons; cancer diagnosis and/or treatment in the last 3 years.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Retention of study participants | 8 weeks
  To estimate retention (measured by number attending the 8 week closeout visit) of men and women being treated for hypertension in the 8 week study.
Adherence to consuming walnuts and EVOO | 8 weeks
  To assess adherence to consuming the nut and oil supplements (measured by daily diary of supplement intake) over the course of the study.

SECONDARY OUTCOMES:
Blood pressure | 8 weeks
  To estimate the variability of blood pressure in men and women participating in the study
Weight | 8 weeks
  To estimate the variability of weight in men and women participating in the study
HDL cholesterol | 8 weeks
  To estimate the variability of HDL cholesterol in men and women participating in the study
Adverse events | 8 weeks
  To document the types and the rates of adverse events associated with the supplements.

CONTACTS AND LOCATIONS:
Overall Officials: Mara Z Vitolins, DrPH MPH RDN, Principal Investigator — Wake Forest University Health Sciences

IPD SHARING:
Plan to Share IPD: No